CLINICAL TRIAL: NCT00316940
Title: A Phase I Study of Samarium Sm-153 Lexidronam Combined With Bortezomib for Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Samarium 153 and Bortezomib in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000479712; ONCOTHER-20051780; ONCOTHER-424Sm35; CYTOGEN-ONCOTHER-20051780
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-12

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; samarium Sm-153 lexidronam

INTERVENTIONS:
Drug: bortezomib
Radiation: samarium Sm 153 lexidronam pentasodium

SUMMARY:
RATIONALE: Radioactive substances, such as samarium 153, may release radiation as it breaks down and kill cancer cells. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Bortezomib may also make tumor cells more sensitive to radiation. Giving samarium 153 together with bortezomib may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of samarium 153 when given together with bortezomib in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety and tolerability (maximum tolerated dose and dose-limiting toxicity) of samarium Sm 153 lexidronam pentasodium and bortezomib in patients with relapsed or refractory multiple myeloma.

Secondary

* Determine the response rate (combined complete response, partial response, and minimal response) in patients treated with this regimen.
* Determine the time to response and the time to progression of disease in patients treated with this regimen.
* Determine the progression-free survival and overall survival of patients treated with this regimen.
* Assess the antitumor effects of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation study of samarium Sm 153 lexidronam pentasodium.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and samarium Sm 153 lexidronam pentasodium IV on day 3. Treatment repeats every 8 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of samarium Sm 153 lexidronam pentasodium until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. The MTD of samarium Sm 153 lexidronam pentasodium is determined with 2 different doses of bortezomib.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with multiple myeloma by 1 of the following criteria:

  * Meets any 2 of the following major criteria:

    * Plasmacytomas on tissue biopsy
    * Bone marrow plasmacytosis (i.e., > 30% plasma cells)
    * Monoclonal immunoglobulin spike IgG > 3.5 g/dL or IgA > 2.0 g/dL by serum electrophoresis; kappa or lambda light chain excretion > 1 g by 24-hour urine protein electrophoresis
  * Plasmacytomas on tissue biopsy AND meets any 1 of the following minor criteria:

    * Presence of monoclonal immunoglobulin at a lesser magnitude than given under above major criteria
    * Lytic bone lesions
    * Normal IgM < 50 mg/dL, IgA < 100 mg/dL, or IgG < 600 mg/dL
  * Monoclonal immunoglobulin spike IgG > 3.5 g/dL or IgA > 2.0 g/dL by serum electrophoresis; kappa or lambda light chain excretion > 1 g by 24-hour urine protein electrophoresis AND meets 1 of the following minor criteria:

    * Bone marrow plasmacytosis (i.e., 10-30% plasma cells)
    * Lytic bone lesions
  * Presence of monoclonal immunoglobulin at a lesser magnitude than given under major criteria with bone marrow plasmacytosis (i.e., 10-30% plasma cells) AND meets 1 of the following minor criteria:

    * Lytic bone lesions
    * Normal IgM < 50 mg/dL, IgA < 100 mg/dL, or IgG < 600 mg/dL
* Measurable disease, defined as a monoclonal immunoglobulin spike of ≥ 1 gm/dL by serum electrophoresis and/or a immunoglobulin spike of ≥ 200 mg by 24-hour urine protein electrophoresis or evidence of lytic bone disease OR
* Nonmeasurable disease (i.e., patients with nonsecretory or oligosecretory multiple myeloma)
* Relapsed or refractory disease

  * Relapsed disease following a response or stable disease after prior chemotherapy (e.g., single-agent steroids, vincristine, doxorubicin, and dexamethasone [VAD], or melphalan and prednisone [MP]) or high-dose chemotherapy
  * Refractory (i.e., failure to achieve at least complete or partial response or stable disease) to the most recent chemotherapy with or without systemic corticosteroids
* No plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein), and skin changes (POEMS syndrome)
* No extramedullary myeloma

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN (unless clearly related to disease)
* Creatinine clearance ≥ 30 mL/min

  * Creatinine clearance > 15 mL/min and < 30 mL/min due to significant myelomatous involvement of kidneys allowed at discretion of investigator
* Sodium > 130 mmol/L
* No ECG evidence of acute ischemia or new conduction system abnormalities
* No myocardial infarction within the past 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No severe hypercalcemia (i.e., serum calcium ≥ 14 mg/dL)
* No New York Hospital Association class III or IV heart failure
* No poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that would preclude study treatment
* No known HIV history
* No known active hepatitis B or C viral infection
* No history of allergic reaction attributable to compounds of similar chemical or biological composition to bortezomib, boron, mannitol, ethylenediaminetetramethylenephosphonic acid (EDTMP), or phosphonates
* No peripheral neuropathy > grade 1

PRIOR CONCURRENT THERAPY:

* At least 12 weeks since prior samarium Sm 153 lexidronam pentasodium

  * No more than 1 prior treatment
* At least 24 weeks since prior strontium chloride Sr 89

  * No more than 1 prior treatment
* No major surgery within the past 4 weeks
* No chemotherapy within the past 3 weeks (6 weeks for nitrosoureas)
* No corticosteroids (> 10 mg/day prednisone or equivalent) within the past 3 weeks
* No immunotherapy, antibody therapy, or radiotherapy (except localized radiotherapy) within the past 4 weeks
* No other concurrent investigational agents
* No concurrent corticosteroids (≥ 10 mg prednisone or equivalent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-12; Primary Completion 2008-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose-limiting toxicity

SECONDARY OUTCOMES:
Response rate (complete, partial, and minimal response)
Time to disease progression and time to response
Progression-free and overall survival
Antitumor effects

CONTACTS AND LOCATIONS:
Overall Officials: James R. Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (4):
- United States (4):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Hematology-Oncology Medical Group of Fresno, Incorporated, Fresno, California
  - West Hollywood, California
  - Center for Cancer and Blood Disorders at Suburban Hospital, Bethesda, Maryland

REFERENCES:
- [Result] Berenson JR, Yellin O, Patel R, Duvivier H, Nassir Y, Mapes R, Abaya CD, Swift RA. A phase I study of samarium lexidronam/bortezomib combination therapy for the treatment of relapsed or refractory multiple myeloma. Clin Cancer Res. 2009 Feb 1;15(3):1069-75. doi: 10.1158/1078-0432.CCR-08-1261. PMID 19188182